CLINICAL TRIAL: NCT01146990
Title: A Prospective, Noninterventional Follow-Up Study of Children Aged 23 to 25 Months, Born to Mothers Who Received Hydroxyprogesterone Caproate Injection, 250 mg/mL, or Vehicle for Prevention of Preterm Birth
Status: Completed | Type: Observational
Sponsor: AMAG Pharmaceuticals, Inc. (Industry)
Collaborators: Registrat-Mapi (Other)
Responsible Party: Sponsor
Other Study IDs: 17P-FU-004
Record Dates: First submitted 2010-06-16; First posted 2010-06-22 (Estimated); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Children Whose Mothers Received 17P and Those Who Received Vehicle in the 17P Efficacy Trial
Keywords: 17P Efficacy Trial Follow up

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Infants Born to Mothers in the 17P-ES-003 Study: Infants Born to Mothers Who Participated in the 17P-ES-003 Study and whose mothers consented for them to be followed for this study.
  Interventions: Drug: ASQ-3, Bayley III, Neurologic exam

INTERVENTIONS:
Drug: ASQ-3, Bayley III, Neurologic exam — Developmental Scales of infant development - Children born to mothers who participated in the 17P-ES-003 study will be enrolled in this study and evaluated using the ASQ-3. Those meeting protocol criteria based on ASQ-3, will be evaluated using the Bayley III and have a neurologic examination.

SUMMARY:
In the continuing efforts to understand the benefits and risks of in utero exposure to 17P this study is designed to evaluate differences in developmental outcomes of children, aged 23 to 25 months, born to mothers who participated in the 17P Efficacy Trial sponsored by Hologic (Protocol number 17P-ES-003).

DETAILED DESCRIPTION:
This will be a prospective, noninterventional follow-up study designed to provide a developmental assessment of children born to mothers who participated in the 17P Efficacy Trial. When subjects reach an age of 23 months after adjustment for gestational age, they will be screened for developmental delay using the 24 month ASQ version 3. Subjects who score positive (fall below the specified cut-off) for developmental delay in 1 or more domains will be referred for the 24 month Bayley Scales of Infant and Toddler Development (3rd edition, Bayley-III) and a neurological examination.

ELIGIBILITY:
Inclusion Criteria:

* 1. Maternal enrollment which resulted in a live birth in the 17P Efficacy Trial: A Multi-center, Randomized, Double-blind Study of Hydroxyprogesterone Caproate Injection, 250 mg/mL, Versus Vehicle for the Prevention of Preterm Birth in Women With a Previous Singleton Spontaneous Preterm Delivery.

  2. During their involvement in the above protocol, mothers must have received at least one dose of study drug (Safety population).

  3. Children between 22 and 25 months of age adjusted for gestational age.

Exclusion Criteria:

* 1. There is no parent/legal guardian available to sign an informed consent. 2. Born to women who are unblinded to study group assignment.

Ages: 22 Months to 25 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children whose mothers received 17P and those who received vehicle in the 17P Efficacy Trial
Sampling Method: Non-Probability Sample
Enrollment: 245 (Actual)
Dates: Start 2010-11-09 (Actual); Primary Completion 2020-08-13 (Actual); Study Completion 2020-08-13 (Actual)

PRIMARY OUTCOMES:
Determine whether there is a difference in developmental status between children whose mothers received 17P and those who received vehicle in the 17P Efficacy Trial | aged 23 to 25 months
  The primary objective of this study is to determine whether there is a difference in developmental status between children, aged 23 to 25 months after adjustment for gestational age, whose mothers received 17P and those who received vehicle in the 17P Efficacy Trial.

CONTACTS AND LOCATIONS:
Locations (40):
- United States (24):
  - Drug Research Analysis Corp, Montgomery, Alabama
  - Watching Over Mothers and Babies Foundation, Tucson, Arizona
  - Grossmont Center for Clinical Research, La Mesa, California
  - Naval Medical Center San Diego, San Diego, California
  - Women's Associates, Colorado Springs, Colorado
  - Tripler Army Medical Center, Honolulu, Hawaii
  - The Women's Clinic, Boise, Idaho
  - Women's Healthcare Associates dba Rosemark WomenCare Specialists, Idaho Falls, Idaho
  - University of Louisville School of Medicine, Louisville, Kentucky
  - Women's Care Physicians/Obstetrical Specialists, PLLC, Louisville, Kentucky
  - Steven Z Lenowitz, MD, LLC, Bel Air, Maryland
  - Saginaw Valley Medical Research Group, LLC/Women's OB GYN, PC, Saginaw, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Lyndhurst Gynecologic Associates, Winston-Salem, North Carolina
  - Triad Research Partners, LLC, Winston-Salem, North Carolina
  - SC Clinical Research Center, LLC, Columbia, South Carolina
  - Women's Physician Group, Memphis, Tennessee
  - Practice Research Organization, Inc., Dallas, Texas
  - Wilford Hall Medical Center, Lackland Air Force Base, Texas
  - Tanner Clinic, Layton, Utah
  - Central Utah Clinic, Division of Mt. Timpanogos Women's Health Care, Pleasant Grove, Utah
  - Salt Lake Women's Center, PC, Sandy City, Utah
  - Naval Medical Center, Portsmouth, Virginia
  - Madigan Army Medical Center, Tacoma, Washington
- Canada (2):
  - The Ottawa Hospital, Ottawa, Ontario
  - Medicine Professional Corporation Obstetrics and Gynaecology, Windsor, Ontario
- Czechia (2):
  - Fakultni nemocnice Hradec Králové, Hradec Králové
  - Fakultní Nemocnice Ostrava, Ostrava
- Hungary (4):
  - Szegedi Tudományegyetem Szülészeti és Nogyógyászati Klinika, Szeged, Csongrád megye
  - Petz Aladár Megyei Oktató Kórház, Győr, Győr-Moson-Sopron
  - Debreceni Egyetem Orvos és Egészségtudományi Centrum, Szülészeti és Nogyógyászati Klinika, Debrecen, Hajdú-Bihar
  - Jósa András Oktatókórház Egészségügyi Szolgáltató Nonprofit Kft., Nyíregyháza, Szabolcs-Szatmár-Bereg
- Russia (3):
  - Kazan State Medical University, Kazan'
  - Krasnoyarsk State Medical University named after Prof. V.F.Voino-Yasenetsky, Krasnoyarsk
  - State Educational Institution Saint Petersburg I.I. Mechnikov State Medical Academy of RosZdrav, Saint Petersburg
- Spain (4):
  - Hospital Vall d'Hebrón, Barcelona
  - Hospital Universitario Puerta Del Mar, Cadiz
  - Hospital Universitario Materno Infantil de Canarias, Las Palmas de Gran Canaria
  - Hospital Universitario La Fe, Servicio de Neonatologia, Valencia
- Institute of Pediatrics, Obstetrics and Gynecology of the Academy of Medical Sciences of Ukraine, Kiev, Ukraine